CLINICAL TRIAL: NCT04121936
Title: The Prevalence of Lower Urinary Tract Symptoms (LUTS) in Poland: Epidemiology of LUTS (Poland LUTS) Study
Brief Title: The Prevalence of Lower Urinary Tract Symptoms (LUTS) in Poland
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Piotr Chlosta (Unknown)
Responsible Party: Principal Investigator, Mikolaj Przydacz, Assistant, Jagiellonian University
Other Study IDs: 1072.6120.160.2019
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: To Evaluate Lower Urinary Tract Symptoms (LUTS) in Poland

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There will be no intervention — There will be no intervention

SUMMARY:
The first large population-based study to evaluate lower urinary tract symptoms (LUTS) in Poland. The study objective is to assess the prevalence and bother of LUTS in the population aged ≥40 years in Poland.

DETAILED DESCRIPTION:
The first large population-based study to evaluate lower urinary tract symptoms (LUTS) in Poland. The study objective is to assess the prevalence and bother of LUTS in the population aged ≥40 years in Poland.

This study will be conducted as a telephone survey with assessment of LUTS using a standardized protocol, which included the International Prostate Symptom Score (IPSS) and, for overactive bladder (OAB), the OAB-V8 questionnaire. Participants will be asked to rate how often they experienced individual LUTS and the degree of associated bother.

The study will be performed in a representative group of Polish population (n = 6,000) covering all geographic regions of Poland (defined by the Central Statistical Office of Poland).

ELIGIBILITY:
Inclusion Criteria:

Age >40

Exclusion Criteria:

Age <40 Pregnancy Urinary tract infection in the past 4 weeks

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative group of Polish population
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of LUTS | Through study completion, an average of 3 months
  The prevalence of LUTS will be assessed using definitions of the International Continence Society (descriptive statistics).
Symptom bother of LUTS | Through study completion, an average of 3 months
  The degree of associated bother will be assessed using Likert scale (Likert scale: not at all [score 0], a little bit [score 1], somewhat [score 2], quite a bit [score 3], a great deal [score 4], or a very great deal [score 5]).

SECONDARY OUTCOMES:
Prevalence of specific symptoms | Through study completion, an average of 3 months
  The prevalence of specific symptoms will be assessed using a standardised protocol based on the definitions provided by the International Continence Society (i.e. storage symptoms, voiding symptoms and post-micturition symptoms) [Abrams P, Cardozo L, Fall M, et al. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21:167-178]. Participants will be asked to rate how often they experienced individual LUTS during the past month. A Likert scale will be used with the following options: none (score 0), <1 in 5 times (score 1), <half the time (score 2), about half the time (score 3), >half the time (score 4), or almost always (score 5).
Symptom bother of specific symptoms | Through study completion, an average of 3 months
  The degree of associated bother of specific symptoms will be assessed using Likert scale (Likert scale: not at all [score 0], a little bit [score 1], somewhat [score 2], quite a bit [score 3], a great deal [score 4], or a very great deal [score 5]).
Prevalence of OAB | Through study completion, an average of 3 months
  The prevalence of OAB will be assessed with the Overactive Bladder-Validated 8-question Screener (OAB-V8)questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology Jagiellonian University, Krakow, Poland

REFERENCES:
- [Derived] Przydacz M, Dudek P, Golabek T, Chlosta P. Relationship between Lower Urinary Tract Symptoms and Treatment-Related Behavior in an Eastern European Country: Findings from the LUTS POLAND Study. Int J Environ Res Public Health. 2021 Jan 18;18(2):785. doi: 10.3390/ijerph18020785. PMID 33477665
- [Derived] Przydacz M, Golabek T, Dudek P, Lipinski M, Chlosta P. Prevalence and bother of lower urinary tract symptoms and overactive bladder in Poland, an Eastern European Study. Sci Rep. 2020 Nov 13;10(1):19819. doi: 10.1038/s41598-020-76846-0. PMID 33188254